CLINICAL TRIAL: NCT01732159
Title: Impact of a Checklist on the Rate of Late Cancellation in Ambulatory Surgery
Acronym: AMBUPROG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: K110601
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Ambulatory Surgery Programmed
Keywords: Ambulatory surgery; Checklist; Cancellation
MeSH Terms: interventions — Checklist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Administration of the checklist (Experimental): Patients will be contacted by phone for administration of the checklist
  Interventions: Other: Checklist
- No contact by phone (No Intervention): Patients who will not be contacted by phone

INTERVENTIONS:
Other: Checklist — he checklist will be administered to the patients by phone between 7 and 3 days before the surgery
  Arms: Administration of the checklist

SUMMARY:
The purpose of this study is to evaluate the impact of a check list on the rate of late cancellation, i.e. the day before or the day of the ambulatory surgery.

DETAILED DESCRIPTION:
The checklist is administered to the patients by phone between 7 and 3 days before the surgery. Each item of the checklist is associated with a decisional algorithm that allows take care for patients in case of any problem.

ELIGIBILITY:
Inclusion Criteria:

* Patient (adult or minor) for which ambulatory surgery is programmed in a multipurpose ASU
* Surgery under general anesthesia or loco
* Regional or neuroleptanalgesia3. Patient contacted by phone
* Patient does not oppose his participation in the study

Exclusion Criteria:

* Patient programmed for endoscopy in ASU non surgical
* Ambulatory surgery scheduled for orthogenic
* Ambulatory surgery scheduled for urgency
* Ambulatory surgery performed under local anesthesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4093 (Actual)
Dates: Start 2012-11; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Decrease in the rate of late cancellation | At day 0 (the day of the surgery)

SECONDARY OUTCOMES:
Improvement of the organization of the ambulatory unit | At day 0 (the day of the surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre BETHOUX, MD, PhD, Principal Investigator — Cochin Hospital
Locations (1):
- Cochin Hospital, Paris, France

REFERENCES:
- [Derived] Gaucher S, Boutron I, Marchand-Maillet F, Baron G, Douard R, Bethoux JP; AMBUPROG Group Investigators. Assessment of a Standardized Pre-Operative Telephone Checklist Designed to Avoid Late Cancellation of Ambulatory Surgery: The AMBUPROG Multicenter Randomized Controlled Trial. PLoS One. 2016 Feb 1;11(2):e0147194. doi: 10.1371/journal.pone.0147194. eCollection 2016. PMID 26829478